CLINICAL TRIAL: NCT06323083
Title: The Effect of Emotional Freedom Technique on Perceived Stress and General Self-Efficacy About Obstetrics and Gynecology Nursing Lesson in Undergraduate Nursing Students With Fear of Birth
Brief Title: The Effect of Emotional Freedom Technique on Perceived Stress and General Self-Efficacy in Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Halime Esra Meram, Principal Investigator, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 006
Record Dates: First submitted 2024-03-14; First posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Emotion Regulation; Stress; Self Efficacy
Keywords: Emotion Regulation; Stress; Self Efficacy; Nursing Student
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Intervention Model Description: The study was designed to be randomly controlled.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Emotional Freedom Technique (EFT) application was applied to those in the intervention group.
  The study was carried out in three stages with three EFT applications, applied for approximately 20-30 minutes, at 7-day intervals. In the first stage, students who met the inclusion criteria were identified by interviewing students who thought they had a fear of childbirth.
  Interventions: Other: Emotional Freedom Technique
- Control group (No Intervention): The control group was also tested at the first interview and again 3 weeks later.

INTERVENTIONS:
Other: Emotional Freedom Technique — Emotional freedom techniques is a psychophysiological intervention that combines psychological methods from traditional therapies with somatic stimulation. EFT involves tapping acupuncture points to desensitize negative emotions by focusing on the emotion.
  Arms: Intervention group

SUMMARY:
The study was conducted to determine the effect of Emotional Freedom Technique (EFT) on perceived stress and general self-efficacy in obstetrics and gynecology nursing lesson in undergraduate nursing students with fear of birth.

The samples were applied to undergraduate nursing students satisfying the research criteria in a state university nursing faculty in Konya at November 2022.

DETAILED DESCRIPTION:
The study was designed to be randomly controlled. Block randomization method was used to determine the intervention and control groups. Randomization was done by a biostatistician outside the researcher. 50 nursing students were randomly assigned to the intervention and control groups. The study was carried out in three stages with three EFT applications, applied for approximately 20-30 minutes, at 7-day intervals. In the first stage, students who met the inclusion criteria were identified by interviewing students who thought they had a fear of childbirth. After informed consent was obtained from the students and pretest data were collected, they were randomly assigned to intervention and control groups. EFT application was applied to those in the intervention group. No intervention was made for the control group. Data was collected twice for the intervention group, before the first EFT application (pretest) and after the last EFT application (posttest). The control group was also tested at the first interview and again 3 weeks later. The applications were carried out face to face with the students as a group. For the collection of research data, "Descriptive Information Form", "General Self-Efficacy (GSE) Scale", "Perceived Stress Scale" and "The Subjective Units of Distress (SUD) Scale" were used.

ELIGIBILITY:
Inclusion Criteria:

* Female students who were taking the Obstetrics and Gynecology Nursing course at the Faculty of Nursing, who volunteered to participate in the study, and who thought they had a fear of childbirth were included in the study.

Exclusion Criteria:

* Female students who did not take the Obstetrics and Gynecology Nursing course at the Faculty of Nursing, did not volunteer to participate in the study, and did not think they had a fear of childbirth were not included in the study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Nursing Students
Enrollment: 50 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2022-11-28 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
General Self-Efficacy Scale | Change from The General Self-Efficacy Scale at three weeks
  The scale consists of 10 items. It is scored between 1-4 and the lowest 10 and the highest 40 points can be obtained.
Perceived Stress Scale | Change from The Perceived Stress Scale at three weeks
  The scale consists of 14 items. It is scored between 0-4 and the lowest 0 and the highest 56 points can be obtained.
The Subjective Units of Distress Scale | Change from The Subjective Units of Distress Scale at three weeks
  It is an 11-point scale commonly used as a subjective verbal rating of discomfort, where 0 indicates absence of discomfort and 10 indicates that it is intolerable.

CONTACTS AND LOCATIONS:
Overall Officials: Halime Esra Meram, PhD, Study Director — Selcuk University
Locations (1):
- Selcuk University, Konya, Turkey (Türkiye)